CLINICAL TRIAL: NCT03086278
Title: A Randomized, Combined SAD/MAD Phase 1 Study of the Safety, Pharmacokinetics and Pharmacodynamics of AST 008 in Healthy Subjects
Brief Title: A Study of AST-008 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Exicure, Inc. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: AST-008-101
Record Dates: First submitted 2017-03-10; First posted 2017-03-22 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Healthy Volunteer Study

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single Ascending Dose (Experimental)
  Interventions: Drug: AST-008

INTERVENTIONS:
Drug: AST-008 — AST-008 is a toll-like receptor 9 agonist.

SUMMARY:
AST-008 will be dosed subcutaneously to healthy volunteers in a combined SAD/MAD study to evaluate its safety, tolerability, pharmacokinetics and pharmacodynamics.

ELIGIBILITY:
Main Inclusion Criteria:

1. Healthy male or female subjects aged ≥18 and ≤40 years of age at the time of first dosing.
2. Subjects must have a body mass index (BMI) between 18.0-25.0 kg/m² inclusive.
3. Satisfactory medical assessment with no clinically significant or relevant abnormalities as determined by medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluation (haematology, biochemistry, coagulation, and urinalysis) that is reasonably likely to interfere with the subject's participation in or ability to complete the study as assessed by the Investigator.
4. Ability to provide written, personally signed, and dated informed consent to participate in the study, in accordance with the ICH Good Clinical Practice (GCP) Guideline E6 (1996) and applicable regulations, before completing any study-related procedures.
5. An understanding, ability, and willingness to fully comply with study procedures and restrictions.

Main Exclusion Criteria:

1. Current or recurrent disease (e.g., cardiovascular, haematological, neurological, endocrine, renal, liver, GI or other conditions) that could affect the action, absorption, or disposition of AST-008, or could affect clinical assessments or clinical laboratory evaluations.
2. Any history of cancer.
3. Any history (including significant and confirmed family history) of autoimmune or antibody-mediated diseases including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, autoimmune hepatitis, or thrombocytopenia.
4. Has had an acute illness within two weeks prior to screening.
5. Current or relevant history of physical or psychiatric illness that may require treatment or make the subject unlikely to fully comply with the requirements of the study or complete the study, or any condition that presents undue risk from the investigational product or study procedures.
6. Any other significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study may influence the result of the study, or the subject's ability to participate in the study.
7. Female subjects who are pregnant or breastfeeding.
8. Subjects with abnormal findings of inguinal, axillary, or cervical lymph nodes at screening or Day -1.
9. A positive human immunodeficiency virus (HIV) antibody screen, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody screen.
10. Titres above reference ranges (according to local laboratory) for autoimmune antibodies: rheumatoid factor (RF), anti-nuclear antibodies (ANA), anti-neutrophil cytoplasmic antibodies (ANCA).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2018-08-16 (Actual)

PRIMARY OUTCOMES:
Serious related adverse events | Up to 1 month after the last dose of AST-008
  To evaluate SAEs after a single subcutaneous dose of AST-008
Adverse events | Up to 1 month after the last dose of AST-008
  To evaluate adverse events after a single subcutaneous dose of AST-008

SECONDARY OUTCOMES:
Dose finding | Up to 1 month after the last dose of AST-008
  To recommend a dose and regimen for further development.
Maximum plasma concentration assessment | Up to 1 month after the last dose of AST-008
  Measurement of the maximum observed plasma concentration (Cmax) after single doses of AST-008
AUC assessment | Up to 1 month after the last dose of AST-008
  Measurement of the area under the curve (AUC) after single doses of AST-008
Pharmacodynamics | Up to 1 month after the last dose of AST-008
  Measurement of type 1 cytokine concentrations as a function of time after single doses of AST-008
Pharmacodynamics | Up to 1 month after the last dose of AST-008
  Measurement of changes in absolute number and and fraction of a panel of lymphocyte markers as a function of time after single doses of AST-008
QTc interval testing | Up to 1 month after the last dose of AST-008
  To determine the effect of AST-008 on QTc interval

CONTACTS AND LOCATIONS:
Locations (1):
- Richmond Pharmacology, London, United Kingdom

REFERENCES:
- [Derived] Daniel WL, Lorch U, Mix S, Bexon AS. A first-in-human phase 1 study of cavrotolimod, a TLR9 agonist spherical nucleic acid, in healthy participants: Evidence of immune activation. Front Immunol. 2022 Dec 13;13:1073777. doi: 10.3389/fimmu.2022.1073777. eCollection 2022. PMID 36582243